CLINICAL TRIAL: NCT05149053
Title: Efficacy of Hydrolyzed Collagen as a Food Supplement in the Reduction of Osteoarticular Pain and Functional Limitation: Results From a Randomized, Double-blind, Placebo-Controlled Study
Brief Title: Hydrolyzed Collagen in the Reduction of Osteoarticular Pain and Functional Limitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francisco Jose Rodriguez Velasco (Other)
Collaborators: NutraResearch, SL (Unknown)
Responsible Party: Sponsor-Investigator, Francisco Jose Rodriguez Velasco, Professor, Universidad de Extremadura
Organization: Universidad de Extremadura (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20/11/2019 CREC
Record Dates: First submitted 2021-11-05; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Osteoarthritis
Keywords: Hydrolyzed Collagen; Osteoarticular Pain; Functional Limitation
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food Supplement (Experimental): Food supplement packet taken one per day preferably in the morning for 6 months.
  Interventions: Dietary Supplement: Hydrolyzed Collagen
- Control (Placebo Comparator): Placebo packet taken one per day preferably in the morning for 6 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Hydrolyzed Collagen — Active product was composed of Hydrolyzed Collagen, lemon flavoring, anhydrous citric acid (acidifier), calcium ascorbate (vitamin C), sucralose (sweetener) and stevia (sweetener). One 10.728 g dose provides 10 g of HC and 80 mg of vitamin C.
  Arms: Food Supplement
Other: Placebo — Placebo packet contained sucralose (sweetener) and stevia (sweetener) in identical proportions to the active preparation.
  Arms: Control

SUMMARY:
This randomised study evaluates the efficacy of an oral dietary supplement of Hydrolyzed Collagen in reducing pain and improving physical function in subjects with osteoarthritis.

DETAILED DESCRIPTION:
In recent years, research efforts have focused on interventions such as collagen supplementation as an alternative treatment for pain and physical function in patients with osteoarthritis. Hydrolyzed collagen (HC) is a mixture of collagen peptides with a molecular weight of less than 5,000 Da. It is obtained from the gelatinization and subsequent enzymatic hydrolysis of native collagen from animal tissues rich in this protein. In this line, several studies show that HC is more easily absorbed enzymatically, has a higher bioavailability, is distributed to joint tissues, and has analgesic and anti-inflammatory properties, consistently showing symptom-relieving effects, thus improving joint function and reducing joint pain, as well as optimizing the patient's quality of life. In this randomized pilot study, the investigators aimed to evaluate the effect on pain and other parameters related to physical function of an oral dietary HC supplement composed of lemon flavoring, anhydrous citric acid (acidifier), calcium ascorbate (vitamin C), sucralose (sweetener) and stevia (sweetener). A 10.728 g dose provides 10 g of HC and 80 mg of vitamin C. Each placebo packet contained sucralose (sweetener) and stevia (sweetener) in identical proportions to the active preparation. Both the active and the placebo were manufactured by NutraResearch© SL (Barcelona, Spain) under Good Manufacturing Practices (GMPs).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of osteoarthritis according to the clinical and radiographic criteria of the American College of Rheumatology.
* Pain score of at a minimum of 50 mm on a VAS scale of 0-100 mm

Exclusion Criteria:

* Presence of a previous cardiovascular event in the last 6 months.
* History of liver or kidney disease.
* Presence of medical condition requiring chronic treatment with drugs or other substances.
* Excessive alcohol consumption (> 20 g/day) or substance abuse.
* Presence of intolerance or hypersensitivity to the food supplement or to any of its components in isolation.
* Use of any intra-articular injection in the anatomical area under study in the last 6 months.
* Treatment with symptomatic slow-acting osteoarthritis drugs (SYSADOA) in the last 3 months.
* Criteria listed in the Clinical Investigation Guideline for medicinal products used in the treatment of osteoarthritis published by the European Medicines Agency of the European Union in 2010 and radiographic osteoarthritis grade 4 according to the Kellgren-Lawrence classification system.
* Any condition that, in the opinion of the investigators, would disqualify the subject from participation in the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Change in baseline osteoarticular pain at 6 months | 0 and 6 months
  Pain level, assessed by Visual Analogue Scale through a repeated measures analysis at two time points (baseline and end of intervention).
Change in baseline functional limitation at 6 months | 0 and 6 months
  Functional limitation, assessed by Lesquene Algofunctional Index through a repeated measures analysis at two time points (baseline and end of intervention)

SECONDARY OUTCOMES:
Change in C-reactive protein (CRP) | 0 and 6 months
  Fasting serum levels of C-reactive protein (CRP), assessed by repeated measures analysis at two timepoints ((baseline and end of intervention).
Change in erythrocyte sedimentation rate (ESR) | 0 and 6 months
  Fasting serum levels of erythrocyte sedimentation rate (ESR), assessed by repeated measures analysis at two timepoints ((baseline and end of intervention).
Patient satisfaction with treatment | 6 months
  Rated with a 3 categories (Good, Poor, Fair), assessed at the end of the intervention.
Treatment-emergent adverse effects | 6 months
  Incidence of adverse effects (type and number) and relatedness to study product (using a 5 category system: certain, likely related, possibly related, conditionally related, unknown), as documented according to the Spanish Medicine and Medical Device Agency (AEMPS) pharmacovigilance system.

CONTACTS AND LOCATIONS:
Locations (1):
- NutraResearch, SL, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No